CLINICAL TRIAL: NCT03385421
Title: Nutritional Practices and Outcomes in Non-Invasive Ventilation
Acronym: NPO-NIV
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, EssaiClinique_NPO-NIV, principal investigator, physician, University Hospital, Grenoble
Other Study IDs: 38RC17.173
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Non Invasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Nutritional Practices and Outcomes in Non-Invasive Ventilation (NPO/NIV) study is a collaboration with lead sites from pediatric critical care units within US and Canada, and participating sites from multiple international regions. The goal of NPO/NIV is to understand how non-invasive ventilation (NIV) is used to treat critically ill children and, concurrently, how these children are fed while on NIV. Designed as a period prevalence study, NPO/NIV will collect observational, cross-sectional data over the course of five study weeks. Each study week will require two days of screening for eligible patients. On Mondays, study staff will screen for patients eligible in the previous 48 hours. On Tuesdays, study staff will screen for patients eligible in the previous 24 hours. Patients meeting study inclusion will be eligible to complete V0, V1, and V2. Included patients will be followed for 7 days after the initiation of NIV or until the patient is discharged from the pediatric intensive care unit. This study was granted exempt status by the University of Arizona Human Subjects Protection Program, including a waiver of informed consent. As no personal health information is transmitted during the course of the study, the University of Arizona does not require Data Use Agreements between sites to participate.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the Pediatric ICU
* in whom noninvasive ventilation (NIV) was initiated within previous 48 hours (NIV use includes any High Flow Nasal Canula > 2 lpm flow , continuous positive airway pressure or bilevel pressure or neurally adjusted ventilatory assist)

Exclusion Criteria:

Patients with:

* chronic home NIV use for >12 hours per day
* limitations of care decisions made
* Cardiac surgery during this admission
* Acute gastro intestinal bleeds
* Abdominal surgery in previous 48 hours
* Gut graft versus host disease
* Chronic parenteral nutrition
* Short Gut Syndrome

Ages: 3 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Population admitted to PICU in whom NIV was initiated
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
hospital mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Katri Typpo, Principal Investigator — University of Arizona
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France